CLINICAL TRIAL: NCT07126912
Title: A Single-arm, Before- After Clinical Study to Evaluate the Safety and Efficacy of Alcarisa Hyaluronic Acid Filler (Espad Pharmed Co.) for Restoration of Mid-face Volume
Brief Title: Evaluation of Efficacy and Safety of Alcarisa (Hyaluronic Acid Produced by Espad Pharmed Co.) for Restoration of Mid-face Volume
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Espad Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALC.ESP.AF.IV.03
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-07

CONDITIONS: Mid Face Volume Deficit

STUDY DESIGN:
Intervention Model Description: before/after clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcarisa (hyaluronic acid filler, produced by Espad Pharmed Co.) (Experimental): A single injection of Alcarisa filler with a maximum dose of 2 to 4 cc , was administered in the zygomaticomalar area, and if deemed appropriate by the physician, also in the anteromedial cheek and submalar areas on each side of the face.
  Interventions: Device: Alcarisa (hyaluronic acid filler)

INTERVENTIONS:
Device: Alcarisa (hyaluronic acid filler) — A single injection of Alcarisa filler with a maximum dose of 2 to 4 cc , was administered in the zygomaticomalar area, and if deemed appropriate by the physician, also in the anteromedial cheek and submalar areas on each side of the face.

SUMMARY:
Mid-face volume loss is a factor affecting beauty that makes people feel uncomfortable about themselves. The purpose of this study is to evaluate the efficacy and safety of Hyaluronic Acid injection with the brand name Alcarisa®, manufactured by Espad Pharmed Co., for treatment of this condition.

The intervention consisted of a single treatment session, injecting 2 to 4 cc of gel into the zygomaticomalar area, and, if deemed by the physician, into the anteromedial cheek and submalar areas on each side of the face.

The patient underwent digital photography at the following time points: before injection, immediately after injection, and at 4, 12, and 24 weeks post-injection. The physician then used these photographs to evaluate the product's efficacy and safety based on predefined measurements. In addition, participant satisfaction was assessed at the same time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 30 to 65 years
* Individuals with moderate to significant mid-face volume loss (score 3 to 4) based on changes in MFVDS (in cases of asymmetry between the two sides of the face, the more severe side will be considered)
* Ability to comply with visit schedules and study procedures
* Signed the informed consent form and agreed to 6-month follow-up

Exclusion Criteria:

* History of Type I hypersensitivity reactions or anaphylaxis
* Known allergy or sensitivity to any components of the filler, lidocaine, or to proteins from the HA-producing microorganisms (Streptococci)
* History of hypertrophic or keloid scarring, or bleeding disorders in the injection area
* Active inflammatory processes, infections, lesions (malignant or benign), or scars in the injection area
* History of streptococcal diseases (such as recurrent sore throat or acute rheumatic fever) in the past 6 months
* History of autoimmune/immunodeficiency diseases, or use of immunosuppressive drugs during the 6 months prior to or during the study
* History of surgery or trauma in the injection area within the past 6 months
* Use of antiplatelet drugs within 72 hours prior to treatment, or anticoagulants within 2 weeks prior to or during treatment
* Use of drugs that reduce or inhibit hepatic metabolism (e.g., cimetidine, beta-blockers) due to the presence of lidocaine
* Pregnancy, breastfeeding, or plans to become pregnant in the near future during the study
* Undergoing or planning to undergo cosmetic treatments in the near future during the study, such as:

  1. Botulinum toxin type A injections below the zygomatic arch during the 6 months prior to study entry
  2. Previous injections of temporary dermal fillers (e.g., bovine collagen, hyaluronic acid) in the facial area within 1 year prior to study entry
  3. Use of calcium hydroxyapatite, poly-L-lactic acid, or permanent fillers (e.g., silicone), or fat injections in the injection area at any time before or during the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
At least one-grade reduction in Midface volume deficit scale (MFVDS) | Baseline, 4 weeks after injection
  At least a one-grade reduction from baseline in Midface volume deficit scale (MFVDS), as assessed by an independent physician based on photographs, where 0 represents no volume deficit and 5 represents severe volume deficit

SECONDARY OUTCOMES:
At least a one-grade reduction in Midface volume deficit scale (MFVDS) | Baseline, 12 and 24 weeks after injection
  At least a one-grade reduction from baseline in Midface volume deficit scale (MFVDS) as assessed by an independent physician based on photographs, where 0 represents no volume deficit and 5 represents severe volume deficit
Depth of the right and left nasolabial folds | 4,12, and 24 weeks after injection
  Depth of the right and left nasolabial folds, measured using standard frontal facial photographs taken with the Visioface device and analyzed via CSI software
Surface area of the right and left nasolabial folds | 4,12, and 24 weeks after injection
  Surface area of the right and left nasolabial folds, measured using standard frontal facial photographs taken with the Visioface device and analyzed via CSI software
Volume of the right and left nasolabial folds | 4,12, and 24 weeks after injection
  Volume of the right and left nasolabial folds, measured using standard frontal facial photographs taken with the Visioface device and analyzed via CSI software
Pain severity during injection | Intervention (day 0)
  evaluated using the Visual Analogue Scale (VAS) from 0 to 10, where 0 indicates no pain at all and 10 indicates the maximum imaginable pain
Participants satisfaction | at 4, 12, and 24 weeks after injection
  Participants' satisfaction assessed using the Visual Analogue Scale (VAS) from 0 to 10, where 0 represents complete dissatisfaction and 10 represents complete satisfaction
Assessment of midface area improvement | at 4, 12, and 24 weeks after the injection
  Assessment of midface area improvement, based on the Global Aesthetic Improvement Scale (GAIS) as judged by the investigator compared to baseline, where 0 means the condition has been worsened and 4 represents excellent improvement
Safety assessment by evaluation of adverse events (AEs) | Immediately after injection; 4, 12, and 24 weeks after injection
  All observed or reported adverse events immediately after injection, as well as 4, 12, and 24 weeks after injection, should be mentioned along with the severity grade (mild = 1, moderate = 2, and severe = 3).

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Center for Research and Training in Skin Disease and Leprocy, Tehran, Tehran Province
  - Orchid Pharmed, Medical Department, Tehran, Tehran Province

IPD SHARING:
Plan to Share IPD: No